CLINICAL TRIAL: NCT04327856
Title: The Assessment of Types and Intensity of Unpleasant Experiences Pre-, Intra-, and Postoperatively in the Patients Undergoing Cataract Surgery, Using Especially Designed Questionnaire.
Brief Title: The Subjective Pre-, Intra-, and Postoperatively Experiences of Patients Undergoing Cataract Surgery.
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Other Study IDs: 1773
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Patient Satisfaction; Patient Compliance; Patient Engagement
Keywords: cataract surgery; quality of life; patient satisfaction; patient experiences
MeSH Terms: conditions — Patient Satisfaction; Patient Compliance; Patient Participation | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cataract surgery group: Patients which were administrated to the Ophthalmology Clinic Medical University of Bialystok due to scheduled cataract removal surgery
  Interventions: Procedure: Cataract Surgery

INTERVENTIONS:
Procedure: Cataract Surgery — The cataract will be removed from patient's eye and artificial intraocular lens will be implanted

SUMMARY:
Assessment of types and intensity of unpleasant experiences pre-, intra-, and postoperatively in the patients undergoing cataract surgery, using especially designed questionnaire.

Strategic aim: formulation of algorithm and modification of perioperative approach to patient qualified to undergo phacoemulsification procedure.

DETAILED DESCRIPTION:
Untreated cataract - the most common reason for an operation in the world - leads to continual decrease in vision, eventually may be the cause of blindness. This condition always requires surgical intervention that involves phacoemulsification with intraocular lens implantation. The procedure takes short amount of time and is performed using topical anaesthesia. Phacoemulsification can be characterised as highly efficient and safe. Besides that, it is still not free from burdens to the patient: causing increased stress levels and anxiety, discomfort or pain, and other symptoms, as surgery is performed on fully conscious and alert patients. Despite, there's lots of research concentrating on patient's quality of life, with different health conditions, the subject of patient's experiences during cataract surgery hasn't been yet fully investigated and explored.

The aim of the study will be an assessment of types and intensity of unpleasant experiences pre-, intra-, and postoperatively in the patients undergoing cataract surgery, using especially designed questionnaire.

Strategic aim: formulation of algorithm and modification of perioperative approach to patient qualified to undergo phacoemulsification procedure.

The prospective questionnaire data will be collected for 200 adults: women and men, that were qualified for cataract surgery in Ophthalmology Department of the Białystok University Clinical Hospital, as an elective surgery with patients being qualified based on specific qualifying criteria.

Based on the questionnaire, that have 128 detailed questions, sociodemographic characteristic of patients will be created, and they will be divided into two groups (I and II) depending whether they are undergoing first or second eye surgery. Juxtaposition of different patients experiences and sensations, with their sociodemographic characteristics, as an implication, will lead to identification of factors that cause surgical procedure to be described either as positive or negative experience. The questionnaire is facilitated also selection of the most significant and frequent reasons for dissatisfaction.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for inclusion required non complicated cataracts (NC1, NC2) according to The Lens Opacities Classification System III (LOCS III scale). Additional inclusion criteria were as follows: documented progression of best corrected visual acuity less than 0.6 according to Snellen notification
* patient agreement to participate in the study after informing them about the nature of the research

Exclusion Criteria:

* bilateral deafness that prevented any communication with the patient;
* no logical contact with the patient (mental disorders, senile dementia, etc.);
* any conditions that might complicate the surgery: post-inflammatory or post-traumatic cataract, chronic corneal disease and corneal opacity that prevent intraoperative vision, advanced disease macular degenerative, active inflammatory process, pregnancy, general steroid therapy.
* lack of patient consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the minimum age of 18, qualified for a routine cataract surgery in Ophthalmology Clinic Medical Univesristy of Bialystok, without any coexisting conditions that might complicate cataract suregery. They were patients of various ages and general health, undergoing first or second cataract surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
The intensity of unpleasant experiences pre-, intra-, and postoperatively | 3 hours post operation
  Assessment of types and intensity of unpleasant experiences pre-, intra-, and postoperatively in the patients undergoing cataract surgery, using especially designed questionnaire.

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Medical University, Bialystok
  - Ophthalmology Clinic Medical University of Bialystok, Bialystok

IPD SHARING:
Plan to Share IPD: Undecided
Individual participants data may be share except any personal details that can enable to make identifiable people who take part in the research i.e. names, surnames, personal identical number

REFERENCES:
- [Background] Lundstrom M, Pesudovs K. Catquest-9SF patient outcomes questionnaire: nine-item short-form Rasch-scaled revision of the Catquest questionnaire. J Cataract Refract Surg. 2009 Mar;35(3):504-13. doi: 10.1016/j.jcrs.2008.11.038. PMID 19251145
- [Background] Friedman DS, Tielsch JM, Vitale S, Bass EB, Schein OD, Steinberg EP. VF-14 item specific responses in patients undergoing first eye cataract surgery: can the length of the VF-14 be reduced? Br J Ophthalmol. 2002 Aug;86(8):885-91. doi: 10.1136/bjo.86.8.885. PMID 12140210
- [Background] Lundstrom M, Roos P, Jensen S, Fregell G. Catquest questionnaire for use in cataract surgery care: description, validity, and reliability. J Cataract Refract Surg. 1997 Oct;23(8):1226-36. doi: 10.1016/s0886-3350(97)80321-5. PMID 9368170
- [Derived] Obuchowska I, Lugowska D, Mariak Z, Konopinska J. Subjective Opinions of Patients About Step-by-Step Cataract Surgery Preparation. Clin Ophthalmol. 2021 Feb 24;15:713-721. doi: 10.2147/OPTH.S298876. eCollection 2021. PMID 33658752
- [Derived] Lugowska D, Konopinska J, Mariak Z, Obuchowska I. Comparison of Subjective Preoperative Experiences of Patients Before First- or Second-Eye Cataract Surgeries. Clin Ophthalmol. 2020 Sep 25;14:2883-2889. doi: 10.2147/OPTH.S270196. eCollection 2020. PMID 33061274